CLINICAL TRIAL: NCT05679934
Title: The Effects of Home-Based Exercise Program And Telerehabilitation on Gait Characteristics, Balance, and Performance in Patients With Normal Pressure Hydrocephalus Applied With Lumbar Puncture
Brief Title: The Effects of Exercise on Gait Characteristics, Balance, and Performance in Patients With Normal Pressure Hydrocephalus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, ümit yeşil, research asistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: deu-uyesil-001
Record Dates: First submitted 2022-12-17; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: NPH (Normal Pressure Hydrocephalus)
Keywords: balance; gait; performance
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-Based Exercise (Experimental): Patients who perform home-based exercise program
  Interventions: Other: Exercise Program
- Telerehabilitation (Experimental): Patients who perform telerehabilitation exercise program
  Interventions: Other: Exercise Program
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Exercise Program — Stretching and strengthening exercises will be applied to the participants
  Arms: Home-Based Exercise; Telerehabilitation

SUMMARY:
The goal of this study is to investigate effect of exercise program on balance, gait and performance in patients with normal pressure hydrocephalus applied with lumbar puncture. The main question it aims to answer are:

* Home based exercise program effective on balance, gait and performance
* Telerehabilitation exercise program effective on balance, gait and performance Researchers will compare home based exercise group, telerehabilitation group and control group to see if difference in terms of balance, gait and performance

ELIGIBILITY:
Inclusion Criteria:

* Age 60-90 years old
* Fulfilling the following clinical criteria for iNPH, as proposed by the Relkin and colleagues
* Able to walk independently (without physical assistance from a person and/or a device)

Exclusion Criteria:

* Patients who had severe physical disability or immobility, major primary psychiatric disorders (eg, schizophrenia, bipolar disorder), unstable major medical illnesses (eg, acute coronary syndrome, respiratory failure), acute cerebrovascular disease, severe visual or hearing impairments were excluded.
* Patients with diagnosis of seconder normal pressure hydrocephalus were also excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Postural Stability | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  Biodex Balance System was used to measure balance-related variables. Biodex has a fixable and movable platform and a touch screen on which the participant can visually track his/her movements.The Postural Stability test emphasizes a patient's ability to maintain center of balance. The device measures anterior-posterior (AP) and medial-lateral (ML) oscillations of the participant and provides anterior-posterior index, medial-lateral index and total stability index scores. Since these scores assess deviations from center, a lower score is more desirable than a higher score
Fall Risk | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  Biodex Balance System was used to measure balance-related variables.Fall Risk test measures the patient's postural sway velocity to predict risk. There is a circular platform that moves freely and simultaneously about the anterior-posterior and medial-lateral axes and provides overall stabiliy index score. The index of overall stability is measured in degrees and higher scores indicate poor dynamic balance
Modified Clinical Test of Sensory Integration of Balance | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  Biodex Balance System was used to measure balance-related variables. mCTSIB provides a generalized assessment of how well patient can integrate various senses with respect to balance and compensate when one or more of those senses are compromised. mCTSIB was performed in four different conditions: eyes open-firm surface (EO-firm), eyes closed-firm surface (EC-firm), eyes open-foam surface (EO- foam), eyes closed-foam surface (EC-foam). The device computes an overall sway index as the standard deviation of the recorded position away from the center. Higher sway index scores indicate greater deviations from the center, therefore, lower scores reflect better response
Walking Speed | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The gait characteristics was measured using G-Walk sensor system. The BTS G-Walk (G-Sensor 2) is a portable, wireless, inertial system with wearable sensors. Each participant was asked to walk down a hallway through a central 7- meter "testing" zone, instructed to walk at his/her ordinary comfortable walking speed and return start line. The acquired data is transmitted via a Bluetooth connection to a computer and processed using the special software program BTS G-Studio.
Cadence | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The test will perform with G-walk device.
Stride Length | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The test will perform with G-walk device.
Time Up and Go Test | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The test will perform with G-walk device.
The Functional Independence Measure | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Functional Independence Measure (FIM) is an assessment tool that aims to evaluate the functional status of patients.FIM is an 18-item, clinician reported scale that assesses an individuals functional capability in six areas including self-care, continence, mobility, transfers, communication and cognition.
Muscle Strength | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  We measured knee extensor and ankle dorsi flexor muscle strength using a hand-held dynamometer. Participants were asked to seat on a bedside (height 100 cm) with hip and knee at 90 degree flexion. Three measurements were taken for each muscle group and the highest score was recorded in kg.

SECONDARY OUTCOMES:
Mini-mental state | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment
The Montreal Cognitive Assessment (MoCA) | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment.
The Clinical Dementia Rating | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Clinical Dementia Rating or CDR is a numeric scale used to quantify the severity of symptoms of dementia
The Geriatric Depression Scale | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly.
The Cornell Scale for Depression in Dementia (CSDD) | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Cornell Scale for Depression in Dementia (CSDD) was specifically developed to assess signs and symptoms of major depression in demented patients.
The Barthel scale | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL).
The Lawton-Brody Instrumental Activities of Daily Living (iADL) | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Lawton-Brody Instrumental Activities of Daily Living (iADL) scale covers eight functional domains: using the telephone, shopping, food preparation, housekeeping, laundry, transport, medication, and finances.
The Tinetti-test | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Tinetti-test, also called Performance-Oriented Mobility Assessment (POMA) assesses a person's perception of balance and stability during activities of daily living and their fear of falling.
The Nine-Hole Peg Test | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses
Grip strength | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength
Fried frailty scale | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  Fried frailty scale is the very first and most commonly used assessment scale for an operational definition of physical frailty with its demonstrated success as a predictor of mobility limitations and mortality. Fried frailty scale includes five components, among which three or more were defined as frailty: unintentional weight loss (10 lbs in the past year), self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity.
FRAIL scale | Change from Baseline at 24 hours after lumbar puncture, change from Baseline at 10 weeks, change from baseline at 24 weeks
  FRAIL scale consists of 5 items; fatigue state, resistance, mobility, weight loss, and existing diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chunyan L, Rongrong H, Youping W, Hongliang L, Qiong Y, Xing L, Yan X. Gait characteristics and effects of the cerebrospinal fluid tap test in probable idiopathic normal pressure hydrocephalus. Clin Neurol Neurosurg. 2021 Nov;210:106952. doi: 10.1016/j.clineuro.2021.106952. Epub 2021 Sep 20. PMID 34619648
- [Background] Hakim S, Adams RD. The special clinical problem of symptomatic hydrocephalus with normal cerebrospinal fluid pressure. Observations on cerebrospinal fluid hydrodynamics. J Neurol Sci. 1965 Jul-Aug;2(4):307-27. doi: 10.1016/0022-510x(65)90016-x. No abstract available. PMID 5889177
- [Background] Gallagher R, Marquez J, Osmotherly P. Gait and Balance Measures Can Identify Change From a Cerebrospinal Fluid Tap Test in Idiopathic Normal Pressure Hydrocephalus. Arch Phys Med Rehabil. 2018 Nov;99(11):2244-2250. doi: 10.1016/j.apmr.2018.03.018. Epub 2018 Apr 25. PMID 29702069
- [Background] Song M, Lieberman A, Fife T, Nielsen M, Hayden S, Sabbagh M, Shi J. A prospective study on gait dominant normal pressure hydrocephalus. Acta Neurol Scand. 2019 Apr;139(4):389-394. doi: 10.1111/ane.13064. Epub 2019 Feb 19. PMID 30676642
- [Background] Schniepp R, Trabold R, Romagna A, Akrami F, Hesselbarth K, Wuehr M, Peraud A, Brandt T, Dieterich M, Jahn K. Walking assessment after lumbar puncture in normal-pressure hydrocephalus: a delayed improvement over 3 days. J Neurosurg. 2017 Jan;126(1):148-157. doi: 10.3171/2015.12.JNS151663. Epub 2016 Mar 18. PMID 26991388
- [Background] Bottcher N, Bremova T, Feil K, Heinze C, Schniepp R, Strupp M. Normal pressure hydrocephalus: Increase of utricular input in responders to spinal tap test. Clin Neurophysiol. 2016 May;127(5):2294-301. doi: 10.1016/j.clinph.2016.01.027. Epub 2016 Feb 28. PMID 27072102
- [Background] Son M, Cheon SM, Youm C, Kim JW. Turning reveals the characteristics of gait freezing better than walking forward and backward in Parkinson's disease. Gait Posture. 2022 May;94:131-137. doi: 10.1016/j.gaitpost.2022.03.009. Epub 2022 Mar 16. PMID 35306381
- [Background] Bovonsunthonchai S, Witthiwej T, Ngamsombat C, Sathornsumetee S, Vachalathiti R, Muangpaisan W, Hengsomboon P, Thong-On S, Jankhum S, Yangyoo P. Effect of spinal tap test on the performance of sit-to-stand, walking, and turning in patients with idiopathic normal pressure hydrocephalus. Nagoya J Med Sci. 2018 Feb;80(1):53-60. doi: 10.18999/nagjms.80.1.53. PMID 29581614
- [Background] Andren K, Wikkelso C, Tisell M, Hellstrom P. Natural course of idiopathic normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2014 Jul;85(7):806-10. doi: 10.1136/jnnp-2013-306117. Epub 2013 Nov 29. PMID 24292998
- [Background] Isik AT, Kaya D, Ates Bulut E, Dokuzlar O, Soysal P. The Outcomes Of Serial Cerebrospinal Fluid Removal In Elderly Patients With Idiopathic Normal Pressure Hydrocephalus. Clin Interv Aging. 2019 Nov 19;14:2063-2069. doi: 10.2147/CIA.S228257. eCollection 2019. PMID 31819388
- [Background] Tisell M, Tullberg M, Hellstrom P, Edsbagge M, Hogfeldt M, Wikkelso C. Shunt surgery in patients with hydrocephalus and white matter changes. J Neurosurg. 2011 May;114(5):1432-8. doi: 10.3171/2010.11.JNS10967. Epub 2011 Jan 14. PMID 21235310
- [Background] Relkin N, Marmarou A, Klinge P, Bergsneider M, Black PM. Diagnosing idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S4-16; discussion ii-v. doi: 10.1227/01.neu.0000168185.29659.c5. PMID 16160425
- [Background] Viteckova S, Horakova H, Polakova K, Krupicka R, Ruzicka E, Brozova H. Agreement between the GAITRite(R) System and the Wearable Sensor BTS G-Walk(R) for measurement of gait parameters in healthy adults and Parkinson's disease patients. PeerJ. 2020 May 22;8:e8835. doi: 10.7717/peerj.8835. eCollection 2020. PMID 32509441
- [Background] Sherafat S, Salavati M, Ebrahimi Takamjani I, Akhbari B, Mohammadirad S, Mazaheri M, Negahban H. Intrasession and intersession reliability of postural control in participants with and without nonspecific low back pain using the Biodex Balance System. J Manipulative Physiol Ther. 2013 Feb;36(2):111-8. doi: 10.1016/j.jmpt.2012.12.005. PMID 23499146
- [Background] Prometti P, Olivares A, Gaia G, Bonometti G, Comini L, Scalvini S. Biodex Fall Risk Assessment in the Elderly With Ataxia: A New Age-Dependent Derived Index in Rehabilitation: An Observational Study. Medicine (Baltimore). 2016 Mar;95(10):e2977. doi: 10.1097/MD.0000000000002977. PMID 26962804
- [Background] Lim TS, Yong SW, Moon SY. Repetitive lumbar punctures as treatment for normal pressure hydrocephalus. Eur Neurol. 2009;62(5):293-7. doi: 10.1159/000235808. Epub 2009 Aug 27. PMID 19713705
- [Background] Rossi PD, Damanti S, Nani C, Pluderi M, Bertani G, Mari D, Cesari M, Consonni D, Spagnoli D. Repeated Cerebrospinal Fluid Removal Procedure in Older Patients With Idiopathic Normal Pressure Hydrocephalus Ineligible for Surgical Treatment. J Am Med Dir Assoc. 2019 Mar;20(3):373-376.e3. doi: 10.1016/j.jamda.2018.11.014. Epub 2019 Jan 9. PMID 30638833
- [Background] Larsson J, Israelsson H, Eklund A, Lundin-Olsson L, Malm J. Falls and Fear of Falling in Shunted Idiopathic Normal Pressure Hydrocephalus-The Idiopathic Normal Pressure Hydrocephalus Comorbidity and Risk Factors Associated With Hydrocephalus Study. Neurosurgery. 2021 Jun 15;89(1):122-128. doi: 10.1093/neuros/nyab094. PMID 33830219
- [Background] Nikaido Y, Kajimoto Y, Akisue T, Urakami H, Kawami Y, Kuroda K, Ohno H, Saura R. Dynamic Balance Measurements Can Differentiate Patients Who Fall From Patients Who Do Not Fall in Patients With Idiopathic Normal Pressure Hydrocephalus. Arch Phys Med Rehabil. 2019 Aug;100(8):1458-1466. doi: 10.1016/j.apmr.2019.01.008. Epub 2019 Feb 4. PMID 30731067
- [Background] Nikaido Y, Urakami H, Okada Y, Kajimoto Y, Ishida N, Kawami Y, Akisue T, Saura R. Dynamic gait stability in patients with idiopathic normal pressure hydrocephalus with high and low fall-risk. Clin Biomech (Bristol). 2022 Oct;99:105757. doi: 10.1016/j.clinbiomech.2022.105757. Epub 2022 Sep 5. PMID 36113194
- [Background] Abram K, Bohne S, Bublak P, Karvouniari P, Klingner CM, Witte OW, Guntinas-Lichius O, Axer H. The Effect of Spinal Tap Test on Different Sensory Modalities of Postural Stability in Idiopathic Normal Pressure Hydrocephalus. Dement Geriatr Cogn Dis Extra. 2016 Sep 27;6(3):447-457. doi: 10.1159/000450602. eCollection 2016 Sep-Dec. PMID 27790243
- [Background] Lundin F, Ledin T, Wikkelso C, Leijon G. Postural function in idiopathic normal pressure hydrocephalus before and after shunt surgery: a controlled study using computerized dynamic posturography (EquiTest). Clin Neurol Neurosurg. 2013 Sep;115(9):1626-31. doi: 10.1016/j.clineuro.2013.02.015. Epub 2013 Mar 11. PMID 23489444
- [Background] Hess T, Milani TL, Meixensberger J, Krause M. Postural performance and plantar cutaneous vibration perception in patients with idiopathic normal pressure hydrocephalus. Heliyon. 2020 Dec 31;7(1):e05811. doi: 10.1016/j.heliyon.2020.e05811. eCollection 2021 Jan. PMID 33458441
- [Background] Ishikawa M, Yamada S, Yamamoto K. Early and delayed assessments of quantitative gait measures to improve the tap test as a predictor of shunt effectiveness in idiopathic normal pressure hydrocephalus. Fluids Barriers CNS. 2016 Nov 22;13(1):20. doi: 10.1186/s12987-016-0044-z. PMID 27876063